CLINICAL TRIAL: NCT01387529
Title: Reference Values for Non-invasive Hydration Status Markers
Brief Title: Reference Values for Non-invasive Hydration Status Markers H10-14
Status: Completed | Type: Observational
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: S-11-15
Record Dates: First submitted 2011-06-30; First posted 2011-07-04 (Estimated); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Value Orientation
Keywords: Reference Values

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The objective of this study is to establish reference values for non-invasive hydration status markers. Although there are no hypotheses associated with this study, the outcome will help advance the development of non-invasive hydration status monitors (described above and in H08-12; A-15208) capable of detecting dehydration from a single, static measure. The outcome that this research effort supports what is recognized by the military community as a high priority medical technology gap (MOM ICD v1.3, 2008).

DETAILED DESCRIPTION:
Disorders of fluid and electrolyte balance in the U.S. military result in at least 125 hospitalizations, two lost duty days per event, and 9,300 ambulatory hospital visits per year (60% hyponatremia, 40% dehydration) (Carter et al., 2005; DoD, 2008). Diarrhea is a major infectious disease threat which requires aggressive i.v. fluid replacement in 30% of U.S. troops deployed to Iraq or Afghanistan (Brown et al., 2009). It is also important to recognize that the management and outcome of the 662 severe or penetrating traumatic brain injuries (TBI) reported for the military in 2009 (DoD, 2010) may be hindered by dehydration (Clifton et al., 2002). Fluid and electrolyte imbalances also contribute to heat illness (Carter et al., 2005) and can substantially impair combat fighting effectiveness (Dupont, 2003).

The importance of developing a valid assessment measure of human hydration status for clinical and field use is recognized by the military community as a high priority medical technology gap (MOM ICD v1.3, 2008). In far forward locations (levels I-II), orthostatic testing or gross symptoms are most commonly used to estimate hydration status (Manning et al., 2007). However, level I-II methods share symptoms with numerous other maladies and are insensitive until dehydration is severe or becomes debilitating (Levitt et al., 1992; McGee, 1999). Definitive hydration assessment in rear roles of medical care (levels III-V) requires invasive serial blood and/or urine measurements (Feig, 1977; Mange, 1997). Thus, a field-expedient technology that provides an accurate, non-invasive assessment of hydration status would improve medical triage by allowing better fluid-electrolyte management by medics in theatre (point of care), and by medical personnel in the rear levels of care (treatment and return to duty).

ELIGIBILITY:
Inclusion Criteria:

* male or female subject over the age of 18 years
* subject in good general health
* written informed consent for participation in the study
* report any adverse events?
* if female of child bearing potential, has the subject confirmed that she is not pregnant
* if the subject wears contact lenses, is he/she willing to remove them

Exclusion Criteria:

* Presence of a significant medical condition, which in the opinion of the investigator precludes participation in the study
* Use of ANY medication other than oral contraceptives

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Approximately 150 volunteers (military and civilians) will complete this experiment. A sample size of 120 volunteers is recommended for characterizing a sample reference population and constructing reference intervals (Fraser, 2001). A sample size of 150 will allow for the potential loss of data due to equipment or handling errors, and 'bad' samples resulting from volunteer non-compliance. A subset of as many as 50 volunteers will undergo repeat testing (3 days; ~3 hours) for the purpose of determining within-subject variance.
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2011-06; Primary Completion 2013-03 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Cheuvront, Ph.D., Principal Investigator — US Army Insititute of Environmental Medicine Thermal & Mountain Medicine Div.
Locations (1):
- US Army Research Institute of Environmental medicine Thermal and Mountain Meidicine Division, Natick, Massachusetts, United States